CLINICAL TRIAL: NCT02136641
Title: Study of Comparison of the Effectiveness of Three Diagrams for Sedation in Spinal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Cartagena (Other)
Responsible Party: Principal Investigator, FRANCISCO JOSE BERMUDEZ GUERRERO, Specialist in Anesthesiology, Universidad de Cartagena
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NCT01651989; p-2011-1682 (Other Grant/Funding Number: Colciencias)
Record Dates: First submitted 2014-05-03; First posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Anesthesia; Reaction
Keywords: Anesthesia; Spinal Anesthesia; Conscious Sedation; Operating Rooms.
MeSH Terms: interventions — Midazolam; Fentanyl; Ketamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Midazolam (Active Comparator): 1. Sedation with Midazolam 0.03 mg / kg, Intravenous, administered as a single dose. Was given to those patients randomly assigned to this group, who were scheduled for procedures previously defined in the inclusion criteria.
  Interventions: Drug: Midazolam
- Midazolam+Fentanyl Combination (Experimental): 2. Sedation with Midazolam 0.015 mg / Kg + Fentanyl 0.8mcg/kg, Intravenous, administered as a single dose. Was given to those patients randomly assigned to this group, who were scheduled for procedures previously defined in the inclusion criteria.
  Interventions: Drug: Midazolam+Fentanyl Combination
- Midazolam+Ketamine Combination (Experimental): 3. Sedation with Midazolam 0,015 mg / Kg + ketamine 0.25 mg / kg, Intravenous, administered as a single dose. Was given to those patients randomly assigned to this group, who were scheduled for procedures previously defined in the inclusion criteria.
  Interventions: Drug: Midazolam+Ketamine Combination

INTERVENTIONS:
Drug: Midazolam — Was applied Midazolam 0.03 mg / kg, IV (in the vein), single dose.
  Arms: Midazolam
Drug: Midazolam+Fentanyl Combination — Was applied Midazolam 0.015 mg / Kg + Fentanyl 0.8mcg/kg, IV (in the vein), single dose.
  Other Names: Midazolam; Fentanyl
  Arms: Midazolam+Fentanyl Combination
Drug: Midazolam+Ketamine Combination — Was applied Midazolam 0,015 mg / Kg + ketamine 0.25 mg / kg, IV (in the vein), single dose.
  Other Names: Midazolam; Ketamine hydrochloride
  Arms: Midazolam+Ketamine Combination

SUMMARY:
Objective: To determine the efficacy of sedation schemes to sedation in patients about to undergo spinal anesthesia.

Methods: Pilot study, clinical type, randomized, prospective, single-blind, in which the investigators compared three schemes for sedation in patients undergoing spinal anesthesia.

Keywords: Anesthesia, Spinal Anesthesia, Conscious Sedation, Operating Rooms.

DETAILED DESCRIPTION:
Sedation is a set of actions aimed at achieving a patient be quiet, comfortable, free of pain and / or bad memories as a diagnostic or therapeutic procedure is performed . Given that regional anesthetic techniques frequently used in clinical practice are relatively traumatic and painful procedures , have partnered on multiple occasions sedation, to make such interventions more comfortable for the patient and make it easier to peer collaboration . Not all anesthesiologists use sedation or indicate similarly, but the vast majority practice it. Some apply it consistently before or after puncture for a regional block or in the event that required multiple punctures, and other used only when the patient is anxious .

There are various drugs for sedation in anesthesiology with multiple anxiolytic, amnesic, and analgesic to, including barbiturates, benzodiazepines, opioid analgesics, and combinations thereof, are proof of this ketamine, midazolam, fentanyl, propofol, dexmedetomidine, and others . There is a clear need to implement sedation techniques that provide effectiveness, safety and few side-effects as well as low cost to search anxiolysis, amnesia, analgesia and / or drowsiness in patients who are undergoing procedures such as spinal anesthesia .

Reducing anxiety and decreased neurological and metabolic response to surgical trauma become a requirement to be treated in the anesthetic plan, sedation there plays a key role in seeking to ensure an adequate hemodynamic stability during locoregional anesthetic techniques under conscious sedation, this being, sedation in which a patient responds normally to verbal stimuli, with preservation of cognitive function and coordination, without alteration of the ventilation or cardiovascular function. The ideal state of sedation depends on the type of patient, type of procedure and the medications used, however it is recommended to maintain a level of sedation between 2 and 3 or conscious sedation, according to Ramsay sedation scale to achieve greater wellness and collaboration, without requiring intervention to keep the airway, while maintaining adequate spontaneous ventilation and cardiovascular function normally held.

The objective is to determine the effectiveness of three sedation schemes in patients scheduled to undergo spinal anesthesia.

MATERIALS AND METHODS A clinical trial, randomized, prospective, single-blind experimental study was conducted, in which three schemes were compared for sedation in patients undergoing spinal anesthesia. Informed consent was obtained from each of the admitted patients. The study was approved by the ethics committee of the University of Cartagena.

Patients who met selection criteria were randomized (according to a table of random numbers generated on the website: http://stattrek.com/tables/random.aspx) to be assigned to one of the research groups, in the period between June 2011 and June 2012.

3 groups were formed as follows: Group 1 was given midazolam 0.03 mg / kg, Group 2 was applied Midazolam 0.015 mg / Kg + Fentanyl 0.8mcg/kg and in Group 3 was used Midazolam 0,015 mg / Kg + ketamine 0.25 mg / kg, administered as a single dose in all groups.

Sample size, with a reliability of 95%, a power of 80% and an expected rate of improvement in experimental group of 80% was calculated , for a total of 75 patients, and were randomly assigned to one of the three study groups, each group consisted of 25 patients. The investigators selected all patients who met the inclusion criteria such as age between 18 and 60 years , scheduled for elective surgery, have pre-anesthetic assessment, be classified according to their risk as ASA I or ASA II, having a body mass index between 18.5 and 29.99, not be pregnant, have a higher fasting 8 hours the day of the procedure, require regional anesthetic technique without contraindications to the procedure and can be performed with the patient in the lateral decubitus , have not known history of allergy, and haven't as an exclusion criteria malformations of the spine level that would prevent a spinal block without difficulty.

Procedure: assigned randomly selected for each patient using a scheme sedation, 75 numbers were randomly through a generator of random number tables , with a minimum value of 1 and a maximum value of 3, and as they selected a patient was applied corresponding scheme in sequential order. On admission to the operating room the patient was channeled to a peripheral vein 18 -20Gauge, were monitored with electrocardiogram (ECG), non -invasive blood pressure (NIBP) and oxygen saturation by pulse oximetry (O2Sat) by a vital signs monitor; hemodynamic variables were recorded income. Was applied intravenously one of the pre-established schemes sedation according to patient weight and oxygen was administered by nasal cannula 1Litre/minutes , hemodynamic changes were recorded at 2.5 and 5 minutes from the scheme were implemented and evaluated the Ramsay scale at the time. The patient is positioned for carrying the anesthetic technique, and with a Quincke needle 26 Gauge, spinal anesthesia by a team of experienced anesthesiology was placed, corresponding to the authors of this study, the number of attempts and difficulty to blockade were noted, at the end of the surgical procedure a satisfaction survey was performed to the patient about their experience with spinal block.

The data collection was performed using a format that included sociodemographic characteristics, variables of interest and two measuring scales were used:

The first was the RANSAY SCALE, which is a scale used to assess the depth of sedation , is validated over 30 years ago, is easy to use and has been the gold standard in many studies that evaluated sedation; as you increase the level on the scale, increasing the degree of sedation . Being awake patient can be found in a level 1, referring to an anxious and / or agitated patients in level 2, when partner is quiet and focused and have spontaneous eye opening, or a level 3 when has closed eyelids, but quickly responds to verbal stimuli. When the patient was found asleep, level 4 will be called if you are still with closed eyes and responds quickly to tactile and verbal stimuli strong, level 5 when it has a slower response and only responds to important and / or painful stimuli and level 6 when does not respond to any stimulus.

In addition, a SATISFACTION SCALE TYPE LIKERT was used to subjectively evaluate how satisfied was the patient with spinal anesthesia under sedation, the scale is not validated , giving a score of 1 to refer to be very satisfied, 2 if only felt satisfied, a score of 3 to be dissatisfied, 4 if it meant feeling unsatisfied and finally a rating of 5 if it meant being very dissatisfied.

Data analysis: the counting of categorical variables are reported as absolute numbers and percentages. Differences in baseline characteristics and post-intervention were estimated through hypothesis testing. For qualitative variables the Chi square test and Fisher's exact test was used, as appropriate. In quantitative variables of normal verified through Shapiro-Wilk test and comparison groups by ANOVA, this analysis was supported with Epi Info v7 and Stata software.

Ethical issues: the declaration of Helsinki and the regulations in force in Colombia (1993 Resolution No.008430 MOH 2378 and resolution 2008 on good clinical practice) was adjusted. No actions against incurring ethical proposals were registered there. Assessment was required by the ethics committee of the Hospital, who gave his endorsement to proceed with its development, a report of individual informed consent of patients was performed.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective surgery
* Have pre-anesthetic assessment
* Be classified according to their risk as ASA I or ASA II
* Having a body mass index between 18.5 and 29.99
* Not be pregnant
* Have a higher fasting 8 hours the day of the procedure
* Require regional anesthetic technique without contraindications to the procedure -Can be performed with the patient in the lateral decubitus
* Have not known history of allergy

Exclusion Criteria:

* Malformations of the spine column level , that creates a lock troubles

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Sedation level reached according RANSAY SCALE with the use of three schemes sedation to spinal anesthesia | one year
  Sedation/Analgesia conscious was considered adequate when a RANSAY 2 or 3 was achieved (BASED ON THE RANSAY SCALE), without the need for other anesthetic drugs are different from the protocol, has been the gold standard in many studies that evaluated sedation; as you increase the level on the scale, increasing the degree of sedation . Being awake patient can be found in a level 1, referring to an anxious and / or agitated patients in level 2, when partner is quiet and focused and have spontaneous eye opening, or a level 3 when has closed eyelids, but quickly responds to verbal stimuli. When the patient was found asleep, level 4 will be called if you are still with closed eyes and responds quickly to tactile and verbal stimuli strong, level 5 when it has a slower response and only responds to important and / or painful stimuli and level 6 when does not respond to any stimulu

SECONDARY OUTCOMES:
Number of participants satisfied with the use of three schemes sedation to spinal anesthesia | one year
  The Satisfaction was measured with a SATISFACTION SCALE TYPE LIKERT, this scale was used to subjectively evaluate how satisfied was the patient with spinal anesthesia under sedation, the scale is not validated, giving a score of 1 to refer to be very satisfied, 2 if only felt satisfied, a score of 3 to be dissatisfied, 4 if it meant feeling unsatisfied and finally a rating of 5 if it meant being very dissatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: FRANCISCO BERMUDEZ GUERRERO, M.D, Principal Investigator — Universidad de Cartagena
Locations (1):
- Universidad de Cartagena, Cartagena, Departamento de Bolívar, Colombia